CLINICAL TRIAL: NCT02362074
Title: Progress at Work - The Impact of Adalimumab on Work Related Productivity in Patients With Rheumatoid Arthritis.
Acronym: P @ Work
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-455
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab subjects: Subjects starting Adalimumab treatment at time of enrollment.

SUMMARY:
The purpose of this study is to describe the impact of treatment with adalimumab on work related productivity and economic burden in patients with Rheumatoid Arthritis (RA) treated in Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with moderate to severe RA for whom the physician has decided to initiate treatment with adalimumab
2. Adult male or female ≥ 18 years old that has been newly prescribed adalimumab therapy according to the local product label and are with PROGRESS
3. Subjects should be evaluated for tuberculosis (TB) exposure/risk factors for active and latent TB
4. Subject is able to give written patient authorization and is willing to comply with the requirements of this study protocol.

Exclusion Criteria:

1. Subject cannot or will not sign a patient authorization
2. Subject with a known hypersensitivity to Adalimumab, or any of its components
3. Presence of any condition that, in the opinion of the treating physician, prohibits the subject from participating in the study or obscures the assessment of the treatment of RA
4. Subjects currently participating in an investigational clinical trial
5. Subjects treated with >1 prior biologic disease-modifying antirheumatic drugs (DMARDs) for RA. Any prior treatment with adalimumab is prohibited
6. Subjects previously treated with targeted synthetic disease modifying agent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a Multi-Center Canadian Observational Study that will enroll rheumatoid arthristis (RA) subjects for whom the treating physician has decided to treat with adalimumab.
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in Rheumatoid Arthritis-Work Instability Scale (RA-WIS) | From Month 0 to Month 6
  This is patient-reported assessment on the impact of adalimumab on the work status of RA patients.
Change in Financial Loss | From Month 0 to Month 6
  This is patient reported assessment of financial burden of RA.

SECONDARY OUTCOMES:
Change in Rheumatoid Arthritis-Work Instability (RA-WIS) | From Month 0 to Month 12, 18 and 24
  This is patient-reported assessment on the impact of adalimumab on the work status of RA patients.
Change in the Financial Loss | From Month 0 to Month 12, 18 and 24
  This is patient reported assessment of financial burden of RA.
Change in patient pain | From Month 0 to Month 24
  Pain is assessed using Visual Analogue Scale (VAS)
Change in Tender Joint Count (TJC) | From Month 0 to Month 24
  This is assessed by the physician.
Change in Disease Activity Score (DAS) 28 | From Month 0 to Month 24
  Disease activity assessment is done by the physician.
Change in patient assessment of Global Disease Activity | From Month 0 to Month 24
  It is assessed using VAS.
Change in Swollen Joint Count (SJC) | From Month 0 to Month 24
  This is assessed by the physician.
Change in physician's assessment of Global Disease Activity | From Month 0 to Month 24
  It is assessed using VAS.
Change in Health Assessment Questionnaire (HAQ) | From Month 0 to Month 24
  This is patient reported functional assessment.
Change in c-reactive protein (CRP)/erythrocyte sedimentation rate (ESR) | From Month 0 to Month 24
  CRP/ESR values are measured as an inflammatory parameter. Low CRP and ESR values mean less inflammation.
Rate of Remission per Disease Activity Scale (DAS) 28 | From Month 0 to Month 24
  The DAS28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 to 10. A DAS28 score less than 2.6 indicates clinical remission.
Rate of Achieving Low Disease Activity (LDA) per Disease Activity Score (DAS) 28 | From Month 0 to Month 24
  The DAS28 is a validated index of rheumatoid arthritis disease activity. Scores range from 0 to 10 with LDA defined as a score from 2.6 to < 3.2.
Rate of Remission Per Clinical Disease Activity Index (CDAI) | From Month 0 to Month 24
  The CDAI is used to evaluate disease activity in patients with Rheumatoid Arthritis.
Rate of Achieving Low Disease Activity (LDA) per CDAI | From Month 0 to Month 24
  The CDAI is a composite index for assessing disease activity. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. LDA was defined as a score from 2.8 to ≤ 10.
Rate of Remission per Simplified Disease Activity Index (SDAI) | From Month 0 to Month 24
  The SDAI is a validated measure of rheumatoid arthritis disease activity. Scores on the SDAI range from 0 to 86 with a SDAI score ≤3.3 indicating clinical remission.
Rate of Achieving Low Disease Activity (LDA) per SDAI | From Month 0 to Month 24
  The SDAI is a validated measure of rheumatoid arthritis disease activity. Scores on the SDAI range from 0 to 86 with a SDAI score <11 indicating LDA.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (32):
- Canada (32):
  - Pont, Cranbrook, BC, CA /ID# 134511, Cranbrook, British Columbia
  - Drs. M & W Teo Inc. /ID# 148641, Penticton, British Columbia
  - The Arthritis Research Center /ID# 147466, Vancouver, British Columbia
  - Kur, Vancouver, CA /ID# 135371, Vancouver, British Columbia
  - Manitoba Clinic /ID# 134830, Winnipeg, Manitoba
  - Nexus Clinical Research /ID# 135411, St. John's, Newfoundland and Labrador
  - St. Clare's Mercy Hospital /ID# 136737, St. John's, Newfoundland and Labrador
  - Dr. Juris Lazovskis Inc. /ID# 134510, Sydney, Nova Scotia
  - Waterside Clinique /ID# 134190, Barrie, Ontario
  - Drs Nalin and Vandana Ahluwali /ID# 136485, Brampton, Ontario
  - Dr. Sanjay Dixit Medicine Professional Corporation /ID# 136486, Burlington, Ontario
  - Dr. Chrisotomor Kouroukis & Dr /ID# 151189, Dundas, Ontario
  - Adachi Medicine Prof. Corp /ID# 152538, Hamilton, Ontario
  - West Mountain Medical Center /ID# 134832, Hamilton, Ontario
  - Dr. Martin M.S. Lee Med Prof C /ID# 138333, Mississauga, Ontario
  - Brandusa Florica Med Prof Corp /ID# 134829, Mississauga, Ontario
  - Montgomery, Mississauga, CA /ID# 136943, Mississauga, Ontario
  - Credit Valley Rheumatology /ID# 134834, Mississauga, Ontario
  - Rajwinder S. Dhillon Medicine /ID# 147756, Niagara Falls, Ontario
  - Capital North Therapeutics Res /ID# 134835, Ottawa, Ontario
  - Setty, Owen Sound, CA /ID# 134189, Owen Sound, Ontario
  - The Medical Centre /ID# 134833, Peterborough, Ontario
  - Involved Medicine /ID# 163880, Toronto, Ontario
  - Dr. Samuel K Silverberg /ID# 136496, Toronto, Ontario
  - Institut de Rhum. de Montreal /ID# 135289, Montreal, Quebec
  - Jewish General Hospital /ID# 204168, Montreal, Quebec
  - PSS Medical Inc. /ID# 134193, Montreal, Quebec
  - Clinique de Rhumatologie de Montréal /ID# 162186, Montreal, Quebec
  - Ctr. de Rheum de l'est du QC /ID# 135410, Rimouski, Quebec
  - Rheum Disease Ctr of Montreal /ID# 135372, Westmount, Quebec
  - Dr. Latha Naik /ID# 135813, Saskatoon, Saskatchewan
  - Chuq - Chul /Id# 137054, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P14-455.pdf